CLINICAL TRIAL: NCT06314217
Title: Everads Injector in Suprachoroidal Administration of a Triamcinolone Acetonide (TA) Suspension Approved for Intraocular Injection, for the Treatment of Patients With Diabetic Macular Edema: An Open-label Safety and Performance Pilot Study
Brief Title: Everads Injector in Suprachoroidal Administration of TA Suspension, for Treatment of Patients With DME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Everads Therapy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CL-00002; 202330714 (Registry Identifier: MOH ISRAEL)
Record Dates: First submitted 2024-03-05; First posted 2024-03-15 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Macular Edema
Keywords: suprachoroidal

STUDY DESIGN:
Intervention Model Description: Everads Injector: For targeted suprachoroidal delivery of therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label prospective device study (Experimental): Treatment of previously treated patients diagnosed with diabetic macular edema (DME)
  Interventions: Device: Everads Injector

INTERVENTIONS:
Device: Everads Injector — Single suprachoroidal injection of triamcinolone acetonide, 4 mg in 100 μl using Everads Injector

SUMMARY:
This is an open-label pilot device study. The aim of the study is to evaluate the safety and performance of Everads Injector following single injection of suspension approved for ocular use into the suprachoroidal space.

The study population is patients diagnosed with diabetic macular edema (DME) that were previously treated. 10 adult subjects are expected to be enrolled based on the inclusion-exclusion criteria.

The study will involve 6 visits during a period of 6 weeks

DETAILED DESCRIPTION:
The study involves 6 visits: Screening Visit: Visit 1 (Day -6 to 0); Baseline and Injection Visit: Visit 2 (Day 1); Follow up visits: Visit 3 (Day 3 ± 1 Days), Visit 4 (Day 14 ± 3 Days), Visit 5 (Day 28 ± 3 Days); End of Trial: Visit 6 (Day 42 ± 3 Days).

Patient eligibility will be assessed at screening, and the study eye will be determined.

Baseline/Injection Visit will include a pre-injection examination, injection of TA and post-injection examination The study eye will receive the suprachoroidal injection of TA injectable suspension approved for ocular use. The Everads Injector will be used for a single administration of 100 µl (4 mg) of TA into the suprachoroidal space in the treatment eye.

Injections using Everads Injector will be performed by trained and qualified investigators after training by Sponsor experts

Study assessments include: physical examination, vital signs, medical & ocular history, AE and concomitant medication assessment.

Ophthalmological examination include:

* Best-corrected visual acuity (BCVA) using the Early Treatment of Diabetic Retinopathy Study (ETDRS) Visual Acuity Chart.
* Intraocular Pressure
* Optical coherence tomography (OCT)
* Fundus photography
* Fluorescein angiography
* ICG angiography
* Slit-lamp biomicroscopy
* Dilated indirect ophthalmoscopy.

Subject will be followed for 42 days following injection

ELIGIBILITY:
Key Inclusion Criteria:

1. Males and females ≥ 18 years of age with a diagnosis of type 1 or type 2 diabetes mellitus.
2. Diagnosis of DME with confirmed central involvement of ≥ 320 µm for males and ≥ 305 µm for females on Spectralis (Heidelberg) or ≥ 305 µm for males and ≥ 290 µm for females with Cirrus (Zeiss) by spectral domain optical coherence tomography (SD-OCT), verified at the screening visit.
3. First three patients: ETDRS BCVA letter score of worse than 35 (Snellen equivalent of 20/200 imperial or 6/60 metric) in the study eye, and ETDRS BCVA of 60 (Snellen equivalent of 20/63 imperial or 6/19 metric) or better in the fellow eye. Remaining patients: ETDRS BCVA letter score of worse than 50 (Snellen equivalent of 20/100 imperial or 6/30 metric) in the study eye, and ETDRS BCVA of 60 (Snellen equivalent of 20/63 imperial or 6/19 metric) or better in the fellow eye.
4. Have shown no response to three previous Intravitreal (IVT) treatments with anti-vascular endothelial growth factor (VEGF) agents.

Key Exclusion Criteria:

1. Evidence of macular edema of any cause other than diabetic retinopathy in the study eye.
2. Prior treatment with pan-retinal photocoagulation or focal laser photocoagulation in the study eye within 90 days of screening visit.
3. Intraocular pressure ≥ 21 mmHg or uncontrolled glaucoma (open-angle or angle-closure) in the study eye.
4. History of any prior ophthalmic surgeries in the study eye within 90 days of the screening visit.
5. Previous treatment for DME in the study eye with any intravitreal injection in the 30 days prior to the screening visit.
6. Any previous treatment with Ozurdex® implant in past 6 months.
7. Any previous treatment with Iluvien® or Retisert™.
8. Current iris neovascularization, vitreous hemorrhage, tractional retinal detachment or epiretinal membrane that contributes to macular edema in the study eye, per PI discretion.
9. Uncontrolled blood pressure.
10. HbA1c >12%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-02-18 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment-emergent adverse events | 6 weeks
  Frequency of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) (6 weeks) TEAEs are defined as events that emerge following administration of TA via the Everads Injector.
Frequency of adverse device effects | 6 weeks
  Frequency of adverse device effects and frequency of serious adverse device effects (SADEs) throughout the study period (6 weeks) Adverse device effects and SADEs are defined as effects that emerge following the use of the Everads Injector.

SECONDARY OUTCOMES:
Confirmation of TA delivery into the suprachoroidal space | Injection day
  Confirmation of TA delivery into the suprachoroidal space, as determined by imaging assessment(s) and/or ocular examination following the injection.
Change from baseline in central macular thickness | 6 weeks
  Change from baseline in central macular thickness (CMT), as measured by OCT.

CONTACTS AND LOCATIONS:
Overall Officials: Barak, MD, Principal Investigator — Rambam MC; Keren Mano Tamir, MD, Study Director — Everads Therapy
Locations (1):
- Rambam MC, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No